CLINICAL TRIAL: NCT04319822
Title: Mobility, Functional Autonomy and Respiratory Function After Prolonged Stay in Intensive Care Unit
Acronym: MAORI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0465_7732
Record Dates: First submitted 2019-06-24; First posted 2020-03-24 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Intensive Care
Keywords: Intensive Care Unit; Prolonged Stay in Intensive Care Unit
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood samples, muscular biopsy, and quality of life (Experimental): quality of life, blood samples, quadriceps biopsy in intensive care unit (before and after the ICU hospitalization and one at M6
  Interventions: Other: blood sample and muscular biopsy

INTERVENTIONS:
Other: blood sample and muscular biopsy — blood sample and muscular biopsy

SUMMARY:
The hospital survival of patients hospitalized after prolonged stay in intensive care unit has improved however there are a loss of functional autonomy and an impaired of peripheral and respiratory muscle performance, what leads to an impairment life's quality. These sequels constitute the Post Intensive Care Syndrome (PICS).

The objective of this cohort is to describe the functional autonomy at 6 months of a prolonged stay in intensive care unit and to study the associations between functional autonomy and 1 / the biological data obtained from quadriceps biopsies / the trajectory of post-resuscitation care.

The primary endpoint is functional autonomy at 6 months of ICU stay, assessed by the Functional Independence Measure (FIM) score.

In order to take into account a rate of loss of sight we propose to include in this cohort 120 subjects during their stay in intensive care unit.

DETAILED DESCRIPTION:
The hospital survival of patients hospitalized after prolonged stay in intensive care unit has improved however there are a loss of functional autonomy and an impaired of peripheral and respiratory muscle performance, what leads to an impairment life's quality. These sequels constitute the Post Intensive Care Syndrome (PICS). Incomplete understanding of the physiopathological mechanisms that allow the recovery of functional autonomy and the lack of consideration of post-intensive care pathway seems central to explain the contrasting results of therapeutic trials in this syndrome.

Incomplete understanding of the physiopathological mechanisms that allow the recovery of functional autonomy and the lack of consideration of post-intensive care pathway seems relevant to explain the contrasting results of therapeutic trials in this syndrome.

The objective of this cohort is to describe the functional autonomy at 6 months of a prolonged stay in intensive care unit and to study the associations between functional autonomy and 1 / the biological data obtained from quadriceps biopsies / the trajectory of post-resuscitation care

Patient at high risk of loss on functional autonomy, staying in the three intensive unit care participants will be recruited, if they present inclusion criteria and don't present exclusion criteria Inclusion criteria: - mechanical ventilation for at least 72 hours and extra-respiratory organ failure Exclusion criteria : neurological or psychiatric deficit preventing the performance of assessment tests, chronic ventilation on tracheotomy, bedridden patient or moribund

The primary endpoint is functional autonomy at 6 months of ICU stay, assessed by the Functional Independence Measure (FIM) score. The secondary endpoints are survival, peripheral and respiratory muscle performance, metabolic stress testing, biologic features associated with muscle regeneration (quadriceps biopsy in resuscitation (before and after) and one at M6) , the quality of life and the path of care post-resuscitation. The statistical analysis will make it possible to describe the population according to 3 groups of the same size according to the Tertiles of the FIM to M6. The analysis will look for variables associated with belonging to the "case" group: patients with the highest disability (last testeile of the FIM score) compared to "controls": patients with a less severe disability (first two tiertiles of the score) FIM). In order to take into account a rate of loss of sight we propose to include in this cohort 120 subjects during their stay in intensive care unit.

Progress: 2 visits are planned (ICU, M6 and monthly telephone interviews). The duration of the inclusions will be 30 months and the duration of the follow-up of the patients will be 6 months.

Prospect :

* identification of physiopathological and structural factors (post-ICU trajectory) associated with recovery of functional autonomy and respiratory and peripheral muscular performance at a distance from a stay in intensive care unit
* the design of a personalized interventional study in order to improve the functional autonomy

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation for at least 72 hours and extra-respiratory organ failure

Exclusion Criteria:

* neurological or psychiatric deficit preventing the performance of assessment tests,
* chronic ventilation on tracheotomy, bedridden patient or moribund

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the functional autonomy of patient | 6 months
  The functional autonomy will be assessed by The Functional Independence Measure test (FIM score) 6 months after ICU

SECONDARY OUTCOMES:
Number of patient survival | 6 months
  Number of alive patient 180 days after stay in intensive care unit
Performance of peripheral and respiratory muscles | 6 months
  Assessment of the patient deambulation assessed by a walking test
metabolic stress testing | 6 months
  Assessment of the metabolic stress testing
Description of the Characterization of satellite cells responsible for muscle regeneration | up to 6 months
  The aim is only to understand and describe the Characterization of satellite cells responsible for muscle regeneration ( PAX -7).
Description of the Biochemical features of the peripheral muscles | up to 6 months
  Global physiological description of the Biochemical features of the peripheral muscles : proteolysis / proteosynthesis balance, mitochondrial fusion / fission markers, autophagy, mitophagy)
Assessment of the patient Quality of life | up to 6 months
  Quality of life assessed by the validated test EQ5D
Assessment of the post ICU medical care and social environement | up to 6 months
  Assessed by the validatedtest : Social Provisions Scale

IPD SHARING:
Plan to Share IPD: Yes
Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 months after the main publication
Access Criteria: Dataset will be shared after careful examination by the study board of investigators.
URL: https://biolincc.nhlbi.nih.gov/studies/